CLINICAL TRIAL: NCT02136472
Title: Female Subfertility: a First Sign of Metabolic and Cardiovascular Anomalies?
Brief Title: Female Subfertility: a Metabolic and Vascular Profile
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Desiree Pattinaja, MD, PhD candidate, Maastricht University Medical Center
Other Study IDs: METC 13-2-001
Record Dates: First submitted 2014-04-30; First posted 2014-05-13 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Metabolic Syndrome X; Infertility
Keywords: Subfertility; Metabolic syndrome; Plasma volume; Intima media thickness; Flow mediated dilatation
MeSH Terms: conditions — Metabolic Syndrome; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subfertile women: Women who visit the fertility clinic of the Maastricht University Medical Centre who start with a basic fertility work-up. Women diagnosed with an unexplained subfertility or with (signs of) a decreased ovarian reserve are asked for further participation in the study of the cardiovascular profile.
  As a control group parous women with an uncomplicated pregnancy more than 6 months ago will be asked for participation.

SUMMARY:
Introduction:

Overall, 10 - 15% of couples seek specialist help once in their lives when a spontaneous pregnancy does not occur. These couples are defined subfertile when there is at least one year of unprotected intercourse without conceiving. Subfertility can have different causes which can be diagnosed with a basic fertility work-up. Unfortunately, the subfertility in 25% of the couples still remains unexplained.

Hypothesis:

The investigators hypothesize that cardio-metabolic and hemodynamic abnormalities reducing cardiovascular reserves relate to circulatory redistribution at the expense of uterine perfusion and with it women's fertility. This could especially be important in the subgroups with an unexplained subfertility and a decreased ovarian reserve. Interventions to improve these abnormalities could lead to better results in fertility treatment, better obstetric outcome and reduced lifelong health risks.

Objective:

The investigators want to examine specific cardio-metabolic and cardiovascular parameters in women of subfertile couples. The investigators want to evaluate the prevalence of metabolic syndrome in all women who are assessed for subfertility compared to healthy parous women. Furthermore in the women with an unexplained subfertility or with (signs of) a decreased ovarian reserve the cardiovascular profile will be studied consisting of the uterine artery pulsatility index (PI) as measure of uterine perfusion, the plasma volume as measure of venous reserve capacity, the intima media thickness of the carotid arteries as proxy of chronic strain and the endothelial function, measured by flow mediated dilatation (FMD) of the brachial artery.

Study design:

Cross-sectional

Study population:

The study group consists of subfertile women between 18 and 41 years who visit the fertility clinic in the Maastricht University Medical Centre with a primary or secondary subfertility. Women with an unexplained subfertility or with (signs of) a decreased ovarian reserve are evaluated for their cardiovascular profile. The control group consists of women with a history of an uneventful spontaneous pregnancy.

Main study parameters:

1. Prevalence of metabolic syndrome in subfertile women
2. The cardiovascular profile, in women with an unexplained subfertility or with (signs of) a decreased ovarian reserve, consisting of:

   * The uterine artery pulsatility index
   * The plasma volume
   * The intima media thickness (IMT)
   * The endothelial function of the vascular system (FMD)

DETAILED DESCRIPTION:
Introduction:

Overall, 10 - 15% of couples seek specialist help once in their lives when a spontaneous pregnancy does not occur. These couples are defined subfertile when there is at least one year of unprotected intercourse without conceiving. Subfertility can have different causes. A basic fertility work-up focuses on the reproductive system of the couple. After this basic fertility work-up the subfertility remains unexplained in 16-24% of the couples. The investigators hypothesize that cardio-metabolic and hemodynamic abnormalities reducing cardiovascular reserves relate to circulatory redistribution at the expense of uterine perfusion and with it women's fertility. This could especially be important in the subgroups with an unexplained subfertility and a decreased ovarian reserve. For all possible assessed abnormalities, proven effective treatments are available such as primarily life style corrective actions. Furthermore these interventions could lead to better results in fertility treatment, better obstetric outcome and reduced lifelong health risks.

Objective:

The overall objective of this study is to examine specific cardio-metabolic and cardiovascular parameters in women of subfertile couples. This study protocol is divided into 3 studies to evaluate several cardio-metabolic/cardiovascular parameters in different subgroups of female subfertility compared to fertile women.

* Study 1 "The metabolic syndrome and female subfertility": The prevalence of metabolic syndrome in all women who are assessed for subfertility compared to fertile women.
* Study 2 "The cardiovascular profile in female subfertility": The cardiovascular profile of women with female subfertility classified as unexplained subfertility or "expected" decreased ovarian reserve compared to fertile women. For this study 4 measurements will be performed: the uterine artery pulsatility index (PI) as measure of uterine perfusion, the plasma volume as measure of venous reserve capacity, the intima media thickness of the carotid arteries as proxy of chronic strain and the endothelial function, measured by flow mediated dilatation (FMD) of the brachial artery.
* Study 3 "The cardiovascular profile of women with a poor ovarian response": The cardiovascular profile of women who had an In Vitro Fertilisation (IVF) population with a "proven" decreased ovarian reserve

With these different studies, the investigators hope to identify possible cardio-metabolic/cardiovascular causes for female subfertility. This can lead to new treatment options for female subfertility, enhancing reproductive and obstetric outcome, and a risk assessment for later in life.

Study design:

We want to perform cross-sectional studies.

Study population:

Study 1:

* Study group: subfertile women between 18 and 41 years who visit the fertility clinic in the Maastricht University Medical Centre with a primary or secondary subfertility, independent of the cause of their subfertility
* Control group: women with a history of an uneventful spontaneous pregnancy

Study 2: Women who finished the basic fertility work up and are diagnosed with:

* an unexplained subfertility: study group 1
* an "expected" decreased ovarian reserve: study group 2 Control group: women with a history of an uneventful spontaneous pregnancy

Study 3: Women who received an IVF treatment in the period of 2010 - 2012 and:

* study group: had a "proven" decreased ovarian response, defined as retrieving 3 oocytes or less at an ovum pick-up, despite maximal ovarian stimulation
* control group: received and IVF/Intracytoplasmic Sperm Injection (ICSI) treatment because of a severe male subfertility

Main study parameters:

Study 1: Prevalence of metabolic syndrome in subfertile women compared to fertile controls.

Study 2: The cardiovascular profile, in women with an unexplained subfertility or an "expected" decreased ovarian reserve, consisting of:

1. The uterine artery pulsatility index as measure for uterine perfusion
2. The plasma volume as measure for venous reserve capacity
3. The intima media thickness (IMT) of the carotid arteries as proxy for chronic strain
4. The endothelial function of the vascular system (FMD)

Study 3: The cardiovascular profile, in women with a poor ovarian response, consisting of:

1. The uterine artery pulsatility index as measure for uterine perfusion
2. The plasma volume as measure for venous reserve capacity
3. The intima media thickness (IMT) of the carotid arteries as proxy for chronic strain
4. The endothelial function of the vascular system (FMD)

ELIGIBILITY:
Inclusion Criteria:

Study 1

* Study group:

  * primary subfertility, defined as having no previous pregnancy, or secondary subfertility, defined as a fertility problem after an ongoing pregnancy
  * age 18 - 41 years
* Control group:

  * women with an uneventful pregnancy in history
  * at least 6 months post partum
  * age 18 - 41 years

Study 2

* Study groups:

  * primary subfertility, defined as having no previous pregnancy, or secondary subfertility, defined as a fertility problem after an ongoing pregnancy
  * age 18 - 41 years
  * participation in study 1
  * no abnormalities in the basic fertility work up ("unexplained subfertility"); study group 1, or "expected" decreased ovarian reserve (Follicle Stimulating Hormone (FSH) > 8 u/l); study group 2
* Control group:

  * women with an uneventful pregnancy in history
  * at least 6 months post partum
  * age 18 - 41 years

Study 3

* Study group:

  * primary subfertility, defined as having no previous pregnancy, or secondary subfertility, defined as a fertility problem after an ongoing pregnancy
  * age 18 - 40 years
  * IVF / ICSI treatment in the period from 2010 - 2012
  * proven decreased ovarian response (≤ 3 oocytes at an ovum-pick up)
  * maximal stimulation dosage of 250 IU FSH per day
* Control group:

  * primary or secondary subfertility
  * age 18 - 40 years
  * IVF / ICSI treatment in the period from 2010 - 2012
  * severe male factor (TMC < 3 million spermatozoa)
  * retrieved ≥ 4 oocytes at an ovum-pick up
  * normal stimulation dosage of 150 IU FSH per day

Exclusion Criteria:

Study 1

* There are no exclusion criteria for the study of the metabolic syndrome in the subfertile study group.
* For the control group exclusion criteria are:

  * current pregnancy
  * hormonal medication
  * breastfeeding

Study 2

For the studies of the measurement of the uterine artery PI, plasma volume, intima media thickness and endothelial function exclusion criteria in all women are:

* hypertension, defined as a blood pressure exceeding 140 mm Hg systolic or 90 mm Hg diastolic, or the use of antihypertensive medication
* diabetes mellitus, defined as a fasting glucose level above 6,1 mmol/L or the use of antidiabetic medication

Additional exclusion criteria for the control group:

* hormonal medication
* current pregnancy
* breastfeeding

Study 3

For the study group as well as the control group exclusion criteria are:

* extirpation of an ovary
* cystectomy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study 1:
  * Study group: subfertile women between 18 and 41 years who visit our fertility clinic in the Maastricht University Medical Centre with a primary or secondary subfertility, independent of the cause of their subfertility
  * Control group: women with a history of an uneventful spontaneous pregnancy
  Study 2: Women who finished the basic fertility work up and are diagnosed with:
  * an unexplained subfertility: study group 1
  * an "expected" decreased ovarian reserve: study group 2 Control group: women with a history of an uneventful spontaneous pregnancy
  Study 3: Women who received an IVF treatment in the period of 2010 - 2012 and:
  * study group: had a "proven" decreased ovarian response, defined as retrieving 3 oocytes or less at an ovum pick-up, despite maximal ovarian stimulation
  * control group: received and IVF/ICSI treatment because of a severe male subfertility
Sampling Method: Probability Sample
Enrollment: 512 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The prevalence of the metabolic syndrome in subfertile women | Within 3 months of start of a basic fertility work-up
  Subfertility is defined as trying to conceive for at least one year but did not lead to a pregnancy.
The cardiovascular profile in subfertile women with an unexplained subfertility or a decreased ovarian reserve | Within 3 months after completing the basic fertility work-up
  The cardiovascular profile consists of the plasma volume as measure of venous reserve, the uterine artery pulsatility index as measure of uterine perfusion, the intima media thickness as proxy of chronic strain and the endothelial function of the vascular system.

CONTACTS AND LOCATIONS:
Overall Officials: Ron JT van Golde, MD, PhD, Principal Investigator — Maastricht University Medical Centre; Marc E Spaanderman, Prof, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands